CLINICAL TRIAL: NCT03393351
Title: Evaluation of a Program for Routine Implementation of Shared Decision-Making in Cancer Care: A Stepped Wedge Cluster Randomized Trial
Brief Title: Implementation of Shared Decision-Making in Cancer Care
Acronym: PREPARED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Isabelle Scholl, Head of Research Group, Prinicipal Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: SCHO 1551/1-2
Record Dates: First submitted 2017-12-19; First posted 2018-01-08 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Cancer
Keywords: Shared Decision-Making; Decision Making; Patient Participation; Patient Centeredness; Health Services Research; Implementation Research; Oncology; Stepped Wedge Design; Mixed Methods
MeSH Terms: conditions — Neoplasms; Patient Participation

STUDY DESIGN:
Intervention Model Description: A stepped wedge design, a variant of the cluster randomized controlled trial feasible to evaluate interventions in routine implementation, will be used. Participating clinics will receive the multifaceted implementation program in a randomized sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared decision-making program (Experimental)
  Interventions: Other: Shared decision-making program
- Usual care (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Shared decision-making program — The intervention is shared decision-making. The implementation strategy to foster shared decision-making in routine cancer care is a multicomponent implementation program. The implementation program consists of the following components:
  1. shared decision-making trainings for health care professionals,
  2. individual coaching for physicians,
  3. patient activation strategy,
  4. provision of patient information material and decision aids,
  5. revision of the clinics quality management documents, and
  6. critical reflection of current organization of multidisciplinary team meetings.
  Implementation: after baseline assessment (t0) for clinic 1, after assessment at t1 for clinic 2, after assessment at t2 for clinic 3.
  Arms: Shared decision-making program
Other: Usual Care — No specific study related intervention. Treatment decisions are made according to current routine practice at the comprehensive cancer center in Germany.
  Arms: Usual care

SUMMARY:
This study aims to evaluate a theoretically and empirically grounded implementation program designed to foster shared decision-making in routine cancer care. The intervention program consists of several components (e.g. training for health care professionals, patient empowerment strategies) that will be rolled out in three clinics at a comprehensive cancer center in Germany.

ELIGIBILITY:
Inclusion Criteria for participating patients:

* diagnosed with neoplasms (ICD 10: C00-D49, excluding D10-D36)
* admitted for inpatient or outpatient treatment at the participating clinics
* age > 18 years
* German-speaking

Exclusion Criteria for participating patients:

* severe cognitive impairment

Inclusion Criteria for participating health care professionals:

* physician or nurse working at the participating clinics

Exclusion Criteria for participating health care professionals:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2131 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in uptake of shared decision-making from the patients' perspective | All clinics: baseline, 8 months, 16 months, 24 months
  Action to employ shared decision-making as measured by the German version of the 9-item Shared Decision Making Questionnaire (SDM-Q-9)

SECONDARY OUTCOMES:
Change in uptake of shared decision-making from external observers' perspective | All clinics: baseline, 8 months, 16 months, 24 months
  Action to employ shared decision-making as measured by the German version of the Observer OPTION 5 scale using audio-recorded medical encounters. The Observer OPTION 5 scale measures the extent to which clinicians involve patients in decision-making. Each of the 5 items is assessed on a scale ranging from 0 to 4 with higher values indicating more involvement of patients in decision-making. A sum score is calculated (ranging from 0 to 20) and rescaled to be between 0 to 100, for ease of interpretation.
Acceptability of shared decision-making from the health care providers' perspective | All clinics: baseline, 8 months, 16 months, 24 months
  Perception that shared decision-making is agreeable, palatable, or satisfactory as measured by an adapted version of the acceptability survey developed by McColl et al.
Readiness for implementing change from the health care professionals' perspective | All clinics: baseline, 8 months, 16 months, 24 months
  As measured by an adapted version of the Organizational Readiness for Implementing Change (ORIC) measure
Appropriateness of shared decision-making from the health care professionals' perspective | All clinics: baseline, 8 months, 16 months, 24 months
  Perceived fit, relevance, or compatibility of shared decision-making for the given practice setting as measured by an adapted version of the IcanSDM measure
Change in penetration of shared decision-making at the clinic level | baseline, 3 years
  Integration of shared decision-making within a setting and its subsystems as measured by routine data from patient experience surveys of the clinics
Change in penetration of shared decision-making in multidisciplinary team meetings | All clinics: baseline, 8 months, 16 months, 24 months
  Integration of shared decision-making within a setting and its subsystems as measured by an adapted version of the Metric for the Observation of Decision Making in Multidisciplinary Team Meetings (MDT-MODe)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Scholl, Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (3):
- Germany (3):
  - University Medical Center Hamburg-Eppendorf, Center for Oncology, II. Medical Clinic and Polyclinic, Hamburg
  - University Medical Center Hamburg-Eppendorf, Center for Surgical Sciences, Department of Gynecology, Hamburg
  - University Medical Center Hamburg-Eppendorf, Head and Neurocenter, Department of Oral and Maxillofacial Surgery, Hamburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scholl I, Hahlweg P, Lindig A, Bokemeyer C, Coym A, Hanken H, Muller V, Smeets R, Witzel I, Kriston L, Harter M. Evaluation of a program for routine implementation of shared decision-making in cancer care: study protocol of a stepped wedge cluster randomized trial. Implement Sci. 2018 Mar 27;13(1):51. doi: 10.1186/s13012-018-0740-y. PMID 29580249
- [Derived] Hahlweg P, Lindig A, Frerichs W, Zill J, Hanken H, Muller V, Peters MC, Scholl I. Major influencing factors on routine implementation of shared decision-making in cancer care: qualitative process evaluation of a stepped-wedge cluster randomized trial. BMC Health Serv Res. 2023 Aug 8;23(1):840. doi: 10.1186/s12913-023-09778-w. PMID 37553560
- [Derived] Scholl I, Hahlweg P, Lindig A, Frerichs W, Zill J, Cords H, Bokemeyer C, Coym A, Schmalfeldt B, Smeets R, Vollkommer T, Witzel I, Harter M, Kriston L. Evaluation of a program for routine implementation of shared decision-making in cancer care: results of a stepped wedge cluster randomized trial. Implement Sci. 2021 Dec 29;16(1):106. doi: 10.1186/s13012-021-01174-4. PMID 34965881